CLINICAL TRIAL: NCT06217406
Title: Preemptive Treatment With Acyclovir in Intubated and Mechanically Ventilated Patients With Herpes Simplex Virus Oropharyngeal Reactivation and One or Less Organ Failure
Brief Title: Preemptive Treatment With Acyclovir in Intubated and Mechanically Ventilated Patients With Herpes (PTH2)
Acronym: PTH2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220800; 2023-505510-26-00 (Other: CTIS)
Record Dates: First submitted 2024-01-03; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Invasive Mechanical Ventilation; HSV Throat Reactivation
Keywords: ICU; invasive mechanical ventilation; HSV; Acyclovir; Preemptive treatment
MeSH Terms: interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACYCLOVIR (Experimental): Intravenous acyclovir (ACYCLOVIR )
  Interventions: Drug: Intravenous acyclovir (ACYCLOVIR )
- PLACEBO (Placebo Comparator): saline bags
  Interventions: Drug: Saline bags

INTERVENTIONS:
Drug: Intravenous acyclovir (ACYCLOVIR ) — Patients randomized in the experimental arm will receive intravenous acyclovir at a dosing of 5 mg/kg/8 hours during 14 days (treatment will be stopped at ICU discharge).
  Arms: ACYCLOVIR
Drug: Saline bags — Patients randomized in the control arm will receive placebo, eg. saline bags (same volume as acyclovir bags) every 8 hours during 14 days (treatment will be stopped in case of ICU discharge).
  Arms: PLACEBO

SUMMARY:
This research aims to assess the interest of preemptive treatment with Acyclovir in mechanically ventilated patients with reactivation of Herpes simplex (HSV) in the throat and failure of one organ or less. HSV reactivation is common in patients hospitalized in an intensive care unit (ICU) on invasive mechanical ventilation. It begins at the oropharyngeal level (incidence up to 20-50%), then progresses downward with contamination of the distal airways (reported incidence of 20-65%). HSV reactivation is associated with high mortality. The investigators aim to disable that, in mechanically ventilated patients with HSV reactivation in the throat and failure of one organ or less, preemptive treatment with Acyclovir may reduce mortality.

To answer the question posed in the research, it is planned to include 246 people hospitalized in intensive care on invasive mechanical ventilation, presenting with HSV reactivation of the throat and one organ failure or less.

DETAILED DESCRIPTION:
Herpes simplex virus (HSV) reactivations are frequent in intensive care unit (ICU) patients receiving invasive mechanical ventilation. HSV reactivation first occurs in the throat (incidence up to 20-50%), then progress through a descending way with HSV reactivation in the lung (incidence reported from 20-65%). In some patients, a true HSV bronchopneumonitis can occur: in a prospective study, Luyt et al. found that 24% of patients ventilated for more than 4 days and having ventilator-associated pneumonia suspicion had HSV bronchopneumonitis. These reactivations have been associated with increased mortality, which could be explained by the virus-induced injury on the lung parenchyma, by the increased rate of bacterial pneumonia associated with viral infection, or by the prolongation of mechanical ventilation induced by the previous factors. However, to date it is still unknown if HSV is really a pathogen with its own morbidity/mortality, or only a bystander (with reactivation occurring preferentially in the most severe patients). The only way to know whether or not HSV reactivation has an attributable mortality is to show that a specific treatment, namely acyclovir, has an impact on mortality. One recent randomized controlled study, the PTH study, found that preemptive acyclovir treatment was not associated with shorter duration of mechanical ventilation, as compared to placebo. However, the 60-day mortality rate of patients having received acyclovir was 22% vs. 33% for patients having received a placebo (delta = 11%, p=0.06). Moreover, in the subgroup of patients with 1 organ failure or less (organ failure being defined as a corresponding organ-SOFA (Sepsis-related Organ Failure Assessment) score of 3 or 4), 60-day mortality was significantly lower in patients receiving acyclovir (9%) than mortality of patients receiving placebo (30%, p =0.004). As mortality was not the primary endpoint of PTH study, these exploratory but promising results have yet to be formally confirmed. Therefore, the investigators aim to demonstrate that, in patients mechanically ventilated with HSV reactivation in the throat and 1 organ failure or less, pre-emptive treatment with acyclovir may decrease mortality.

This study is a multicenter, randomized, double-blind, placebo-controlled, concealed allocation superiority trial of intravenous acyclovir vs. placebo for mechanically ventilated patients with 1 organ failure or less and HSV reactivation in the throat. Patients ventilated >96 hours and without exclusion criteria will be screened twice weekly for HSV reactivation using quantitative PCR on swab collected in the throat.

Patients with HSV reactivation will be included and randomized into 2 groups (1:1): acyclovir or placebo. Patients will receive intravenous acyclovir or placebo during 14 days. To keep the blind design of the study, acyclovir and placebo will be reconstituted and/ diluted before the administration in saline bag by the pharmacy or a research's dedicated person (according to sites' possibilities) and dispensed to clinicians. Study drug will be stopped in patients discharged from ICU before end of treatment, i.e. if the patient is discharged before 14 days post randomization.

Allocation concealment will be centralized using a secure web-based randomization system. Patients will be reviewed daily in ICU, at hospital discharge and/or at day 60 post-randomization. Vital status, nosocomial bacterial and viral infection will be collected from day 1 to ICU discharge or day 60. Vital status will be collected at day 90. If discharged from hospital prior to 90 days, the patient (or substitute decision-maker if unable to communicate) will be contacted by telephone to determine the disposition and vital status.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 year-old
* invasive mechanical ventilation(MV) for 96 hours and planned to last for at least 48 hours longer
* HSV reactivation in the throat (qualitative PCR positive for HSV on a throat swab)
* Presence of 1 or less organ failure; organ failure being defined as a corresponding-organ SOFA score of 3 or 4 (for example, renal failure will be defined as a renal SOFA score of 3 or 4)
* Effective contraception for patients of childbearing age, throughout the treatment period
* Written consent from the patient, from a close relative or from the person of trust previously appointed (or inclusion procedure in emergency situations)
* Under social security cover

Exclusion Criteria:

* Hypersensitivity to acyclovir and excipient
* Pregnant or breastfeeding (controlled by a blood pregnancy test)
* Patient who received an antiviral drug active against HSV (acyclovir, valacyclovir, gancyclovir, valgancyclovir, foscavir, cidofovir) in the previous 30 days
* Duration of ventilation before randomization >15 days
* Neutropenia, defined by an absolute neutrophils count < 1,000/mm3
* Solid organ or bone-marrow transplant
* Immunosuppressive treatment (including steroids at a dose >0.5 mg/kg/day of prednisone or equivalent for >1 month)
* HIV infection
* Moribund, defined by a Simplified Acute Physiology Score (SAPS) II score at inclusion >75 points
* Decision of withholding/withdrawing care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | day 60
  Primary endpoint will be the mortality at day 60 post randomization

SECONDARY OUTCOMES:
Mortality | Vital status at day 90 will be assessed either by visit if the patient is still in the hospital, or by phone is the patient is discharged from the hospital
  Day 90
Duration of mechanical ventilation | from date of randomization until the date of extubation or death, whichever first occurs, up to 60 days
  Duration of mechanical ventilation, either invasive or non-invasive, from randomization to extubation or death, whichever first occurs
Ventilator-free days at day 60 | day 60 post-randomization
  Measured as the number of day alive and without mechanical ventilation (invasive mechanical ventilation or non-invasive mechanical ventilation) from randomization to day 60 post-randomization. Patients dying before day 60 will have zero ventilator-free days.
ICU length of stay | from date of randomization until the date of ICU discharge or death, up to 60 days
  Measured by the number of day in the ICU from randomization to ICU discharge or death
ICU-free days | day 60 post-randomization
  measured as the number of day alive and outside the ICU from randomization to day 60 post-randomization. Patients dying before day 60 will have zero ICU-free days.
Hospital length of stay | from date of randomization until the date of hospital discharge or death, up to 60 days
  Measured by the number of day in the hospital from randomization to hospital discharge or death
Hospital-free days | Day 60 post randomization
  Measured as the number of day alive and outside the hospital from randomization to day 60 post-randomization. Patients dying before day 60 will have zero ICU-free days.
Sepsis-related Organ Failure Assessment (SOFA) score (if patient is still hospitalized in ICU) | at days 1, 3, 5, 7, 10, 14, 21 and 28 post-randomization
  This score will be collected using measures collected routinely in the ICU (clinical parameters, blood sampling) A score of two or more is associated with a 10% mortality risk in patients with suspected infection.
Incidence of HSV oral-labial lesions | Oral-labial lesions suggestive of being due to HSV in patients randomized in the study will be recorded. These lesions will be sampled and samples will be sent to the virology laboratory, looking for HSV using polymerase chain reaction (PCR).
  at day 28
Rate patient wth HSV positive in the throat | at days 3, 7, 10, 14, 17, 21 and 28 post randomization
Rate of patient with HSV positive in the tracheal aspirate (if patient is still hospitalized in ICU) | at days 1, 7, 14, 21 and 28 post randomization
  HSV viral load will be measure by quantitative PCR in tracheal aspirate at all time points. Samples will be centralized and analyzed in the French national reference center for herpesviridae.
Rate of HSV bronchopneumonitis | day 60 post randomization
  HSV bronchopneumonitis will be defined by clinical signs suggestive of pneumonia, and presence of HSV in bronchoalveolar lavage (BAL) with a virus load > 105 copies/ millions of cells, whether or not patient had bacterial-viral (namely HSV and bacteria) co-infection.
Rate of acute respiratory distress syndrome (ARDS) | day 60 post randomization
  ARDS will be defined according to Berlin criteria . Patients mechanically ventilated in the ICU have routinely chest X-ray and blood gases analyses, parameters needed to diagnose ARDS. These parameters collected routinely will be used to define ARDS
Rate of bacterial ventilator-associated pneumonia | day 60 post randomization
  Ventilator-associated pneumonia will be defined as clinical signs suggestive of pneumonia, associated with a positive bacteriological sampling. Episodes of ventilator-associated pneumonia will be collected from randomization to day 60.
Rate of bacteremia | day 60 post randomization
  Bacteremia will be defined as a single positive blood culture for pathogenic bacteria, or 2 different blood culture yielding the same pathogen for saprophytic bacteria. Frequency and source of bacteremia will be recorded
Glasgow coma scale (GCS) (if patient is still hospitalized in ICU) | at days 1, 3, 5, 7, 10, and 14 post-randomization.
  Score range from 3 (completely unresponsive) to 15 (responsive) ; Lower GCS scores are correlated with higher risk of death
Creatinine clearance (if patient is still hospitalized in ICU) | at days 1, 3, 5, 7, 10, 14, 21 and 28 post randomization
Number of patients requiring renal replacement therapy | day 14 post randomization
Renal replacement therapy- free days | day 14 post randomization
  Measured as the number of day alive and without need for renal replacement therapy from randomization to day 14 post-randomization. Patients dying before day 14 will have zero renal replacement therapy-free days
Incidence of adverse event, severe adverse event | at days 1, 3, 5, 7, 10, 14, 21 and 28 post randomization
  Intensity and frequency of adverse event and severe adverse event according to the WHO Toxicity Grading Scale for Determining The Severity of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Edouard LUYT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris